CLINICAL TRIAL: NCT02989025
Title: Progesterone to Enhance the Efficacy and Success of Expectantly Managed Preterm Severe/Superimposed Preeclampsia-The PROGRESS Pilot Study
Brief Title: Progesterone to Enhance the Efficacy and Success of Expectantly Managed Preterm Severe/Superimposed Preeclampsia
Acronym: PROGRESS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Babbette Lamarca, Chair and Professor, Pharmacology and Toxicology, University of Mississippi Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0029
Record Dates: First submitted 2016-11-28; First posted 2016-12-12 (Estimated); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Pregnancy; Preeclampsia (PE)
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Experimental (Experimental): To determine if the addition of 17 OHPC to the management of Severe PE diagnosed prior to 34 weeks gestation improves maternal and perinatal outcomes.
  Interventions: Drug: 17 OHPC
- Control (No Intervention): To determine how close the molecular markers are with 17 OHPC added to the management protocol.

INTERVENTIONS:
Drug: 17 OHPC — The study participant will be given 17 OHPC, 250mg IM at admission and every 7 days thereafter.
  Arms: Experimental

SUMMARY:
The purpose of this study is to learn if giving 17-hydroxyprogesterone caproate (17 OHPC) to mothers with preeclampsia diagnosed before 34 weeks gestation improves mother and baby outcomes.

DETAILED DESCRIPTION:
The OBGYN house and attending staff on duty caring for the patient will determine appropriateness for study inclusion. The treating physician will then immediately contact the MFM fellow on call and Research Division personnel to facilitate the initiation of study procedures, including the consent process and baseline blood tests. Once enrolled with informed consent, the participant will receive 17 OHPC, 250mg IM to be given at admission and every 7 days thereafter. Blood sampling of approximately 1-2 teaspoons each will be collected at baseline immediately prior to administration of 17 OHPC, then 24 hours (+-2hrs). After the first 24 hours, blood samples will be collected every 72 hrs until delivery and again 24hrs (+- 2hrs) after delivery. Placentas will be collected at delivery and the investigators will also collect information of the mother and newborn while in the hospital and until discharge including de-identified routine ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* UMMC antepartum patients with preterm PE between 23 0/7ths and 34 0/7ths weeks gestation when initially evaluated
* Willing and able to understand study procedures and to provide informed consent

Exclusion Criteria:

* >33 weeks gestational age or <23 weeks gestation
* Maternal compromise requiring emergent delivery (ongoing placental abruption, DIC, pulmonary edema).
* Fetal compromise requiring emergent delivery (fetal bradycardia, recurrent late fetal heart rate decelerations, minimal to absent fetal heart rate variability).
* Parameters according to current practice guidelines that exclude a patient from expectant management include the following:
* Preterm premature rupture of membranes (PPROM) > 34 weeks gestation;
* Platelet count < 100,000/microliter (thrombocytopenia) with evidence of HELLP syndrome;
* Persistently abnormal hepatic enzyme concentrations (twice or more upper normal values);
* Severe fetal growth restriction (ultrasound-estimated fetal weight less than fifth percentile);
* Severe Oligohydramnios (AFI < 5cm)
* Reversal of end diastolic flow(REDF) in umbilical artery Doppler testing;
* Recurrent (> 2 readings > 30 minutes apart) severe hypertension despite antihypertensive therapy;
* Eclampsia;
* Pulmonary edema;
* Abruption placentae;
* Nonreassuring fetal status during daily testing (biophysical profile <4/10 and/or recurrent variable or late decelerations);
* IUFD

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female only
Enrollment: 60 (Estimated)
Dates: Start 2017-05-22 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Improvement of maternal and perinatal outcomes | Baseline
  Assessment of maternal BP trends

SECONDARY OUTCOMES:
Change is being assessed in Maternal Outcomes | 24 hours
  Assessment of maternal BP trends

OTHER OUTCOMES:
Change is being assessed in Maternal Outcomes | 48 hours
  Assessment of maternal BP trends
Change is being assessed in Maternal Outcomes | Until delivery
  Assessment of maternal BP trends
Assessment of Placental Abruption | Baseline until delivery
  Assessment of Placental Abruption
Assessment of Pulmonary edema | Change from Baseline until delivery
  Assessment of Pulmonary edema
Assessment of Acute Kidney Injury | Change from Baseline until delivery
  Assessment of Acute Kidney Injury
Assessment of DIC | Change from Baseline until delivery
  Assessment of DIC
Assessment of neurological events | Change from Baseline until delivery
  Assessment of neurological events
Assessment of laboratory results | Change from Baseline until delivery
  Assessment of laboratory results
Assessment of Biomarkers | Change from Baseline until delivery
  Assessment of Biomarkers
Assessment of Infant Weight | Delivery
  Assessment of Infant Weight
Assessment of APGAR score | Delivery
  Assessment of APGAR score
Assessment of NICU stays | Delivery
  Assessment of NICU stays
Assessment of Interventricular hemorrhage | Delivery
  Assessment of Interventricular hemorrhage
Assessment of Respiratory Distress Syndrome | Delivery
  Assessment of Respiratory Distress Syndrome
Assessment of Necrotizing enterocolitis (NEC) | Delivery
  Assessment of Necrotizing enterocolitis (NEC)

CONTACTS AND LOCATIONS:
Overall Officials: Babbette LaMarca, PhD, Principal Investigator — University of Missisippi Medical Center; Sheila S Belk, Study Director — UMMC Pharmacology and Toxicology
Locations (1):
- Winfred L. Wiser Hospital, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No